CLINICAL TRIAL: NCT00930826
Title: Childhood Asthma and Schooling: The Truth Unveiled
Acronym: CAS
Status: Completed | Type: Observational
Sponsor: Boushahri Clinic Medical Center (Other)
Responsible Party: Medical Director, Mohamed Said EL-Sayed
Other Study IDs: 461956
Record Dates: First submitted 2008-12-01; First posted 2009-07-02 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2008-11

CONDITIONS: Bronchial Asthma
Keywords: The effect of bronchial asthma on school performance
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Childhood Asthma and Schooling: The Truth Unveiled.

DETAILED DESCRIPTION:
Children with mild persistent asthma still performed worse than normal healthy children in school. The aim of the study was to evaluate school performance of children with mild persistent asthma in comparison with normal healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bronchial asthma
* Must be able to swallow tablets

Exclusion Criteria:

* Steroid inhalation or ingestion

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Residents of a certain town
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)